CLINICAL TRIAL: NCT05475951
Title: Investigation of Gasdermin-D and Pannexin-1 in Fat and Placental Tissues in Pregnant Women With Obesity
Brief Title: Gasdermin-D and Pannexin-1 in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 95932
Record Dates: First submitted 2022-07-06; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy Complications; Maternal Obesity
Keywords: gasdermin-D; pannexin-1; placenta; omental tissue; fat tissue; maternal obesity; inflammation; oxidative stress; biochemistry; ELISA
MeSH Terms: conditions — Pregnancy Complications; Pregnancy in Obesity; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Weight Pregnant Women (Experimental): The women who had term pregnancy and had normal BMI.
  Interventions: Diagnostic Test: Biomarker measurement of pannexin-1 and gasdermin-D
- Overweight Pregnant Women (Experimental): The women who had term pregnancy and had BMI values between 25-30.
  Interventions: Diagnostic Test: Biomarker measurement of pannexin-1 and gasdermin-D
- Obese Pregnant Women (Experimental): The women who had term pregnancy, and had BMI values more than 30.
  Interventions: Diagnostic Test: Biomarker measurement of pannexin-1 and gasdermin-D

INTERVENTIONS:
Diagnostic Test: Biomarker measurement of pannexin-1 and gasdermin-D — These biomarkers were measured in the placental and adipose tissues of the participants.

SUMMARY:
One -third of fertile women around the world are overweight or obese. This means increasing risk for both the mother and the child. Fat tissue is a factor in gestational DM development and the increase in material inflammation and oxidative stress. According to new knowledge, it is an important need to examine molecules that are not handled in new and human research in these mechanisms in fat and placenta tissues in obesity. For this purpose, the examination of the expression of gasdermin-D and pannex-1 proteins, which are shown to be produced in the cells of both tissues, is worth investigating in human fat tissue and placenta. Gasdermins and pannexins are proteins intersecting by interacting in cellular functions.

Gasdermins cause piroptosis, a type of litic proinflammatory cell death. Pannexin-1 plays in various cellular functions, including inflammation. These are examined in a small number of in vitro studies in material fat tissue and placenta, and the design of this study in people whose applications are applied is original in humans.

The status of the expressions of the gasdermin-D and pannexin-1 proteins, which will be examined for the first time in obese pregnant women's fat and placental tissues, are the subject of this research with each other and their relationship with other maternal and neonatal data.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 20-35 age range
* Term pregnancy (37-41 weeks)
* Healthy pregnancy follow-up
* Planned cesarean section
* Having no complication in cesarean delivery
* Being a placenta with front or rear walls

Exclusion Criteria:

* Intrauterine surgical procedure
* Presence of prenatal placental structural disorder
* Multiple pregnancies

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 79 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Prediction of macrosomy | 7 months
  Prediction of macrosomy will be assesed by meaningfull increases of studied biomarkers Gasdermin-D and Pannexin-1

CONTACTS AND LOCATIONS:
Overall Officials: Ali Cetin, Professor, Study Director — Departmant of Obstetrics and Gynecology in Hasek, Training and Research Hospital, Istanbul, Turkey
Locations (1):
- Haseki Training and Research Hospital, Sultangazi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Estienne A, Bongrani A, Reverchon M, Rame C, Ducluzeau PH, Froment P, Dupont J. Involvement of Novel Adipokines, Chemerin, Visfatin, Resistin and Apelin in Reproductive Functions in Normal and Pathological Conditions in Humans and Animal Models. Int J Mol Sci. 2019 Sep 9;20(18):4431. doi: 10.3390/ijms20184431. PMID 31505789
- [Background] Rancourt RC, Ott R, Ziska T, Schellong K, Melchior K, Henrich W, Plagemann A. Visceral Adipose Tissue Inflammatory Factors (TNF-Alpha, SOCS3) in Gestational Diabetes (GDM): Epigenetics as a Clue in GDM Pathophysiology. Int J Mol Sci. 2020 Jan 12;21(2):479. doi: 10.3390/ijms21020479. PMID 31940889
- [Background] Broz P, Pelegrin P, Shao F. The gasdermins, a protein family executing cell death and inflammation. Nat Rev Immunol. 2020 Mar;20(3):143-157. doi: 10.1038/s41577-019-0228-2. Epub 2019 Nov 5. PMID 31690840
- [Background] Abrahams VM, Tang Z, Mor G, Guller S. NLRP3 inflammasome function and pyroptotic cell death in human placental Hofbauer cells. J Reprod Immunol. 2020 Nov;142:103214. doi: 10.1016/j.jri.2020.103214. Epub 2020 Oct 3. PMID 33152658
- [Background] Zhang C, Zhao C, Chen X, Tao R, Wang S, Meng G, Liu X, Shao C, Su X. Induction of ASC pyroptosis requires gasdermin D or caspase-1/11-dependent mediators and IFNbeta from pyroptotic macrophages. Cell Death Dis. 2020 Jun 18;11(6):470. doi: 10.1038/s41419-020-2664-0. PMID 32555186
- [Background] Dye ZT, Rutledge LV, Penuela S, Dyce PW. Pannexin 1 inhibition delays maturation and improves development of Bos taurus oocytes. J Ovarian Res. 2020 Aug 24;13(1):98. doi: 10.1186/s13048-020-00704-w. PMID 32838805
- [Background] Chen KW, Demarco B, Heilig R, Shkarina K, Boettcher A, Farady CJ, Pelczar P, Broz P. Extrinsic and intrinsic apoptosis activate pannexin-1 to drive NLRP3 inflammasome assembly. EMBO J. 2019 May 15;38(10):e101638. doi: 10.15252/embj.2019101638. Epub 2019 Mar 22. PMID 30902848
- [Background] Korac A, Srdic-Galic B, Kalezic A, Stancic A, Otasevic V, Korac B, Jankovic A. Adipokine signatures of subcutaneous and visceral abdominal fat in normal-weight and obese women with different metabolic profiles. Arch Med Sci. 2021 Feb 26;17(2):323-336. doi: 10.5114/aoms/92118. eCollection 2021. PMID 33747267
- [Background] Stubert J, Reister F, Hartmann S, Janni W. The Risks Associated With Obesity in Pregnancy. Dtsch Arztebl Int. 2018 Apr 20;115(16):276-283. doi: 10.3238/arztebl.2018.0276. PMID 29739495
- [Background] Poston L, Harthoorn LF, Van Der Beek EM; Contributors to the ILSI Europe Workshop. Obesity in pregnancy: implications for the mother and lifelong health of the child. A consensus statement. Pediatr Res. 2011 Feb;69(2):175-80. doi: 10.1203/PDR.0b013e3182055ede. PMID 21076366
- [Result] Tozzi M, Hansen JB, Novak I. Pannexin-1 mediated ATP release in adipocytes is sensitive to glucose and insulin and modulates lipolysis and macrophage migration. Acta Physiol (Oxf). 2020 Feb;228(2):e13360. doi: 10.1111/apha.13360. Epub 2019 Oct 14. PMID 31400255